CLINICAL TRIAL: NCT05197829
Title: Glycemic Optimization On Discharge From the Emergency Room
Acronym: GOOD-ER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mark O'Connor (Other)
Responsible Party: Sponsor-Investigator, Mark O'Connor, Assistant Professor, University of Massachusetts, Worcester
Organization: University of Massachusetts, Worcester (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H00023559
Record Dates: First submitted 2021-12-13; First posted 2022-01-20 (Actual); Results first posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-03

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Continuous Glucose Monitoring (Experimental)
  Interventions: Device: Continuous Glucose Monitoring; Other: Care Coordination
- Care Coordination (Active Comparator)
  Interventions: Other: Care Coordination

INTERVENTIONS:
Device: Continuous Glucose Monitoring — Participants in the experimental arm will receive an unblinded flash continuous glucose monitor.
  Arms: Continuous Glucose Monitoring
Other: Care Coordination — All participants will receive diabetes education, written handouts, and help setting up ambulatory appointments.

SUMMARY:
Continuous glucose monitors can help people with diabetes avoid blood sugar levels that are either dangerously high or low. This study evaluates whether continuous glucose monitoring after discharge from the emergency room can help people with type 1 or type 2 diabetes avoid repeat emergency room visits, achieve improved blood sugar control, and feel less distressed about managing their diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Seen in the Emergency Department for hypo- or hyperglycemia
* Either an existing diabetes center patient or a new referral
* Type 1 or type 2 diabetes
* Able to provide informed consent
* Fluent in English or Spanish

Exclusion Criteria:

* Current CGM use
* Need for hospital admission
* Upcoming CT or MRI within 2 weeks
* Pregnancy
* Altered mental status
* Not appropriate for diabetes center follow up
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2023-01-05 (Actual); Study Completion 2024-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark J O'Connor, MD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- UMass Memorial Medical Center, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual-level data underlying published results will be shared with other researchers at the discretion of the principal investigator in accordance with local and institutional policies.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Continuous Glucose Monitoring | Care Coordination
Started | 16 | 14
Completed | 16 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Continuous Glucose Monitoring | Care Coordination | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Continuous [Mean (Full Range); unit: years] | 56 [30 to 85] | 60 [40 to 88] | 58 [30 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 9 | 9 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 5 | 12
  Not Hispanic or Latino | 9 | 9 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 4 | 10
  White | 9 | 9 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 16 | 14 | 30
Type 2 Diabetes [Count of Participants; unit: Participants] | 15 | 14 | 29
New Diagnosis [Count of Participants; unit: Participants] | 10 | 3 | 13
Baseline A1c [Mean (Standard Deviation); unit: percentage of glycated hemoglobin] | 11.5 (2.6) | 10.6 (3) | 11.1 (2.8)

OUTCOME MEASURES:

1. Primary Outcome: Change in Diabetes Distress
Description: Diabetes-related distress will be measured via the 17-question Diabetes Distress Scale (DDS). A higher score indicates more diabetes-related distress. The scale ranges from 1 (low distress) to 6 (high distress).
Time Frame: Change from emergency room visit to first outpatient follow-up visit (2 or 3 weeks)
Population: We analyzed data for patients who completed both the intake survey and the follow-up survey. Some participants never completed the follow-up survey.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Continuous Glucose Monitoring | Care Coordination
Number analyzed (Participants) | 12 | 10
units on a scale | 0 (1.1) | 0.5 (1)

2. Primary Outcome: Outpatient Clinic Attendance Rate
Description: This outcome will measure whether or not each participant attends a subspecialty follow-up appointment as recommended by the emergency room care team.
Time Frame: Follow-up visits will generally occur within 2 or 3 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous Glucose Monitoring | Care Coordination
Number analyzed (Participants) | 16 | 14
Participants | 12 | 9

3. Primary Outcome: Change in the Problem Areas in Diabetes Score
Description: Each participant will fill out the five-question Problem Areas In Diabetes (PAID5) scale. A higher score indicates worse quality of life. Scores range from 0 (good quality of life) to 20 (poor quality of life).
Time Frame: Change from emergency room visit to first outpatient follow-up visit (2 or 3 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Continuous Glucose Monitoring | Care Coordination
Number analyzed (Participants) | 12 | 10
units on a scale | 0 (5.8) | 2.3 (3.2)

4. Secondary Outcome: Number of Patients With Repeat Emergency Utilization
Description: This metric will include repeat emergency room visits and emergency medical services calls.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous Glucose Monitoring | Care Coordination
Number analyzed (Participants) | 16 | 14
Participants | 5 | 7

5. Secondary Outcome: Change in Hemoglobin A1c
Description: Hemoglobin A1c values drawn as part of routine care will be recorded. A positive value indicates that the hemoglobin A1c was lower at follow up than it was at baseline.
Time Frame: 6 Months
Population: We analyzed data for participants who had both a baseline A1c and a follow-up A1c, regardless of whether they attended clinic follow-up visits or not. Some participants did not have follow-up A1c values and were not included in this analysis.
Measure: Mean (Standard Deviation); unit: percentage of glycated hemoglobin
Arm/Group | Continuous Glucose Monitoring | Care Coordination
Number analyzed (Participants) | 10 | 10
percentage of glycated hemoglobin | 5.2 (3.3) | 2.4 (3.4)

6. Secondary Outcome: Outpatient Visits for Which the CGM Data Changed Management
Description: For each patient in the CGM arm, the provider will complete a survey at the time of the initial outpatient follow-up appointment.
Time Frame: 2-3 Weeks
Population: We analyzed data for all provider surveys received.
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous Glucose Monitoring
Number analyzed (Participants) | 10
Participants | 7

7. Secondary Outcome: Time In Range
Description: For participants in the continuous glucose monitoring arm, we will measure the percentage of time spent with a blood sugar level between 70 and 180 mg/dl.
Time Frame: Up to 14 days after the initial emergency visit
Population: We analyzed data for all participants who wore the CGM and returned to clinic with data.
Measure: Mean (Full Range); unit: Percentage of time
Arm/Group | Continuous Glucose Monitoring
Number analyzed (Participants) | 9
Percentage of time | 37 [0 to 95]

8. Secondary Outcome: Percentage Time CGM Active
Description: For participants in the continuous glucose monitoring arm, we will measure the amount of time the sensor was worn.
Time Frame: Up to 14 days after the initial emergency visit
Population: We analyzed data for all participants who wore the CGM and returned to clinic with data.
Measure: Mean (Full Range); unit: Percentage of time
Arm/Group | Continuous Glucose Monitoring
Number analyzed (Participants) | 9
Percentage of time | 73 [24 to 100]

9. Secondary Outcome: Number of Sensor Checks Per Day
Description: For participants in the continuous glucose monitoring arm, we will measure the number of times per day the sensor was used to check a blood sugar level.
Time Frame: Up to 14 days after the initial emergency visit
Population: We analyzed data for all participants who wore the CGM and returned to clinic with data.
Measure: Mean (Full Range); unit: Scans per day
Arm/Group | Continuous Glucose Monitoring
Number analyzed (Participants) | 9
Scans per day | 15 [1 to 36]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Continuous Glucose Monitoring | Care Coordination
All-Cause Mortality (participants affected / at risk) | 1/16 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14
Other Adverse Events (participants affected / at risk) | 0/16 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-29): https://cdn.clinicaltrials.gov/large-docs/29/NCT05197829/Prot_SAP_000.pdf